CLINICAL TRIAL: NCT02955043
Title: A Pilot Trial of a Biobehavioral Intervention to Enhance Hematopoietic Stem Cell Transplant Recovery
Brief Title: Biobehavioral Intervention to Enhance Hematopoietic Stem Cell Transplant Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW16057; P30CA014520 (NIH); NCI-2016-01508 (Registry Identifier: NCI ID Number); 2016-0914 (Other: Institutional Review Board); K07CA136966 (NIH); 4UL1TR000427-10 (NIH); A538900 (Other: UW Madison); SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison)
Record Dates: First submitted 2016-10-31; First posted 2016-11-04 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-09

CONDITIONS: Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Plasma Cell Myeloma; Lymphoid Leukemia; Myeloid Leukemia; Myelodysplastic Syndromes; Multiple Myeloma
Keywords: Hematopoietic Stem Cell Transplantation (HSCT); Fatigue; Insomnia; Depression; Behavioral Intervention
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma; Leukemia, Lymphoid; Leukemia, Myeloid; Myelodysplastic Syndromes; Fatigue; Sleep Initiation and Maintenance Disorders; Depression | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral intervention (Experimental): Participants will learn behavioral techniques to improve sleep and increase daytime activity with the goal of alleviating insomnia, fatigue, and depression. The intervention will be delivered in three 45-60 minute face-to-face sessions at approximately 3-4, 8, and 12 weeks post-HSCT with brief telephone coaching calls scheduled between sessions. Participants will be encouraged to use the behavioral strategies from hospital discharge through 18 weeks post-HSCT. Participants will be asked to complete a daily checklist indicating which intervention strategies they used. Participants will also receive standard medical care following HSCT.
  Interventions: Behavioral: Behavioral techniques
- Usual care (No Intervention): Participants will receive standard medical care following HSCT.

INTERVENTIONS:
Behavioral: Behavioral techniques — Improve nighttime sleep: Participants will receive a modified form of cognitive-behavioral therapy for insomnia with a primary focus on stimulus control, a set of techniques to strengthen the association between bed and sleep and weaken its association with stimulating behaviors.
  Increase daytime activity: Participants will receive instruction in activity management strategies including prioritizing activities, planning activities during peak energy, activity pacing, and alternating between rest and activity. Participants will be provided with a basic step-count pedometer to enhance ability to self-monitor activity and increase motivation for activity.
  The intervention will be adapted to individual needs based on assessments of sleep and activity patterns.
  Arms: Behavioral intervention

SUMMARY:
The goal of this project is to conduct a pilot randomized clinical trial (RCT) to evaluate the feasibility of a brief, behavioral intervention to improve recovery following hematopoietic stem cell transplantation (HSCT). Cancer patients who were treated with HSCT will learn behavioral techniques to improve sleep and increase daytime activity with the goal of alleviating insomnia, fatigue, and depression. If the intervention demonstrates evidence of feasibility and acceptability, a future study will test the effects in a larger trial, with the long-term goal of improving the care and quality of life of cancer survivors recovering from HSCT.

DETAILED DESCRIPTION:
Hematologic cancer patients undergoing hematopoietic stem cell transplantation (HSCT) frequently experience physical and psychological sequelae that impair their quality of life and undermine recovery. Findings from the investigators' laboratory and others indicate that insomnia, fatigue, and depression are among the most persistent, distressing, and debilitating quality-of-life concerns after HSCT. These symptoms co-occur as a "cluster" among cancer patients. Modifying sleep and circadian rest-activity patterns has been suggested to be a particularly promising intervention strategy for alleviating this symptom cluster. The proposed project will therefore evaluate the feasibility and acceptability of a biobehavioral intervention to alleviate insomnia, fatigue, and depression by optimizing sleep and rest-activity patterns during the first 4 months following HSCT. Evidence-based behavioral strategies to enhance the quality of nighttime sleep and increase engagement in non-sedentary daytime activity will be combined to optimize 24-hour rest-activity patterns. These non-pharmacologic approaches can be taught in a few brief sessions and will be delivered in an individual format tailored to each patient.

The investigators have already refined the intervention based on preliminary feasibility testing in a small sample of HSCT recipients and are now conducting a pilot RCT to compare the refined intervention with usual care among adults recovering from HSCT. Semi-structured interviews will determine participant satisfaction with and acceptability of the intervention. Proposed outcome assessments will also be piloted, including patient-reported fatigue, depression, and insomnia measures and actigraphy assessments. The primary goal is to evaluate the feasibility and acceptability of the intervention. The exploratory goal is to conduct a preliminary test of the efficacy of the intervention to determine estimates of variance and effect sizes for determination of power and sample size for a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing hematopoietic stem cell transplantation (HSCT) at the University of Wisconsin Carbone Cancer Center (UWCCC)
* Autologous transplant recipients with multiple myeloma or lymphoma (both Hodgkin's and Non-Hodgkin's types)
* Allogeneic transplant recipients hospitalized for at least 10 days will also be eligible to participate
* Participants who develop treatment complications or disease recurrence after being enrolled in the study may continue to participate if they are able to do so

Exclusion Criteria:

* Autologous transplant recipients with diagnoses other than multiple myeloma or lymphoma
* Allogeneic transplant recipients hospitalized for less than 10 days (a small proportion of allogeneic transplant recipients at UWCCC) will be excluded.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Ability to recruit patients | At the time eligible patients are approached to explain study, up to 40 minutes
  Ability to recruit patients will be evaluated by tracking percent of eligible patients who provide informed consent to the study.
Ability to recruit patients | At the time eligible patients are approached to explain study, up to 20 minutes
  Ability to recruit patients will be evaluated by examining reasons for non-participation.
Ability to retain participants | 18 weeks post-transplant
  Ability to retain participants will be will be evaluated by tracking retention rates through the 18-week study period.
Ability to collect complete data from participants | 18 weeks post-transplant
  Ability to collect complete data from participants will be evaluated by examining rates of completion of study assessments.
Participant willingness to be randomized and acceptability of the usual care condition | 4 weeks post-transplant
  Participant willingness to be randomized will be evaluated by examining attrition between enrollment and the first intervention session.
Participant willingness to be randomized and acceptability of the usual care condition | 18 weeks post-transplant
  Participant willingness to be randomized and acceptability of the usual care condition will be evaluated by examining responses to a semi-structured interview of usual care participants at 18 weeks post-transplant.
Satisfaction with and acceptability of the behavioral techniques | 18 weeks post-transplant
  Satisfaction with and acceptability of the behavioral techniques will be evaluated by examining participants' responses to a semi-structured interview at 18 weeks post-transplant.
Satisfaction with and acceptability of the behavioral techniques | 18 weeks post-transplant
  Satisfaction with and acceptability of the behavioral techniques will be evaluated by examining scores on the Client Satisfaction Questionnaire (CSQ-8) at 18 weeks post-transplant.
Satisfaction with and acceptability of the behavioral techniques | 12 weeks post-transplant
  To examine intervention uptake, participants will complete daily checklist to indicate which intervention strategies they tried between the initial and final intervention sessions.
Acceptability of the assessment strategy | 18 weeks post-transplant
  Acceptability of the assessment strategy will be evaluated by examining participant responses to a semi-structured interview at 18 weeks post-transplant.
Acceptability of the assessment strategy | 18 weeks post-transplant
  Acceptability of the assessment strategy will be evaluated by examining rates of completion of study assessments.
Validity of the assessment strategy | 18 weeks post-transplant
  To address validity, the ability to predict PROMIS measures with the legacy measures the investigators have previously used successfully with this patient population will be assessed. Strong prediction will imply that the PROMIS measures are a statistically valid approach to quantifying the effects of the intervention.

SECONDARY OUTCOMES:
NIH Patient Reported Outcomes Measurement Information System (PROMIS) Sleep disturbance | Pre-transplant, 9 weeks (mid-intervention) and 18 weeks (post-intervention) post-transplant
  A preliminary test of the efficacy of the intervention will be conducted to determine estimates of variance and effect sizes for determination of power and sample size for a larger trial.
NIH Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue | Pre-transplant, 9 weeks (mid-intervention) and 18 weeks (post-intervention) post-transplant
  A preliminary test of the efficacy of the intervention will be conducted to determine estimates of variance and effect sizes for determination of power and sample size for a larger trial.
NIH Patient Reported Outcomes Measurement Information System (PROMIS) Depression | Pre-transplant, 9 weeks (mid-intervention) and 18 weeks (post-intervention) post-transplant
  A preliminary test of the efficacy of the intervention will be conducted to determine estimates of variance and effect sizes for determination of power and sample size for a larger trial.
Actigraphy indices | Pre-transplant, 9 weeks (mid-intervention) and 18 weeks (post-intervention) post-transplant
  The Actiwatch-2 (Philips Respironics), a wrist-worn actigraphy device, will be used to objectively quantify circadian rest-activity patterns over a continuous 7-day period using 1-minute sampling epochs. A traditional cosinor approach will be applied to yield the following indices: mesor (mean activity level), amplitude (rhythm height), acrophase (time of day the rhythm peaks), and R-squared (goodness-of-fit or robustness of the rhythm). The indices will also be compared to determine the effects of the intervention on rest-activity patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Costanzo, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — http://www.uwhealth.org/uw-carbone-cancer-center/cancer/10252